CLINICAL TRIAL: NCT01388582
Title: The Effect of 30mcg and Levonorgestrel 150 Combined Oral Contraceptive, Etonogestrel-releasing Subdermal Implant and Levonorgestrel-releasing Intrauterine System on Breast-Milk Production and Infant Growth in Fully Breast-Feeding Women
Brief Title: The Effect of Hormonal Contraceptives on Breast-milk Production and Infant Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luis Bahamondes, MD Medical Doctor, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06/2011/PC
Record Dates: First submitted 2011-06-16; First posted 2011-07-06 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Underweight
Keywords: contraceptives; hormonal; breastfeeding; infant weight
MeSH Terms: conditions — Thinness; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combined oral contraceptive (Active Comparator): 10 women will receive COC during breastfeeding
  Interventions: Drug: 30 mcg EE and 150 LNG oral contraceptive (Microvlar); Device: TCu380A intrauterine device
- Levonorgestrel intrauterine system (Active Comparator): 10 women will receive a LNG-IUS during breastfeeding
  Interventions: Device: LNG-IUS; Device: TCu380A intrauterine device
- Implanon (Active Comparator): 10 women will receive Implanon during breastfeeding
  Interventions: Device: Implanon; Device: TCu380A intrauterine device
- TCu380A intrauterine device (Active Comparator): 10 women will receive a TCu380A intrauterine device as non hormonal contraceptive during breastfeeding
  Interventions: Device: TCu380A copper-intrauterine device; Device: TCu380A intrauterine device

INTERVENTIONS:
Device: LNG-IUS — 10 women will receive the LNG-IUS during breastfeeding
  Other Names: Mirena, Bayer, Brazil
  Arms: Levonorgestrel intrauterine system
Device: Implanon — 60 mcg/day contraceptive implant
  Other Names: Implanon, MSD, Brazil
  Arms: Implanon
Drug: 30 mcg EE and 150 LNG oral contraceptive (Microvlar) — 10 women will receive oral contraceptive during breastfeeding
  Other Names: Microvlar (Bayer, Brazil)
  Arms: Combined oral contraceptive
Device: TCu380A copper-intrauterine device — Tcu380A copper-intrauterine device will be inserted on 10 women during breastfeeding as non-hormonal comparator group
  Other Names: Optima IUD (Injeflex, Brazil)
  Arms: TCu380A intrauterine device
Device: TCu380A intrauterine device — 10 women will receive a TCu380A intrauterine device as non hormonal contraceptive method during breastfeeding
  Other Names: Implanon, MSD, Os, The Netherland; Mirena, Bayer Oy, Tuku, Finland; TCu380A copper intrauterine device; Optima, Injeflex, Brazil; Microvlar oral contraceptive, Bayer, São Paulo, Brazil

SUMMARY:
The investigators propose a randomized clinical trial comparing the effect of 30 mcg ethinyl estradiol and LNG 150 combination oral contraceptive pills versus placebo, or LNG-IUS or Etonogestrel-releasing contraceptive implant (Implanon)on breast-milk intake and infant growth in exclusively breastfeeding mother-infant pairs. Mother-infant pairs will be randomly assigned either 30 microgram ethinyl estradiol combination oral contraceptive pills or identical placebo to start on post-partum day number 42 or Implanon implants or a LNG-IUS. All women will be offered nonhormonal contraceptives prior to randomization. The pairs will then be followed for four weeks. During this follow-up period, breast-milk intake will be quantified by administering deuterium oxide to exclusively breast-feeding mothers and measuring the enrichment of deuterium oxide in the saliva of their infants, otherwise known as the dose-to-mother method of Coward.17 Additionally, maternal and infant anthropometric measurements will be collected -- both as a value necessary to implement the breast-milk quantification method, as well as an outcome for analysis, and a daily diary will be kept by the women participating in the study that records infant feeds and diaper changes.

DETAILED DESCRIPTION:
Women where allocated to an oral combined contraceptive pill, or placebo or a LNG-IUS or a etonogestrel-releasing subdermal contraceptive implant at day 42 after delivery. After the provision of the contraceptive method a 0.5 mg/kg of deuterium 99.99% according to the weight of the mother will be administer to all women. One sample of saliva from the mother and the child will be collected every day until 21 days after enrollment. Additionally, weight, height and size of the leg of each child will be measured at baseline, at the day 11 and at the day 21 after enrollment. Also, a diary with information of change of diapers and number of breastfeeding will be kept by each mother.

ELIGIBILITY:
Inclusion Criteria:

* women at the day 42th of post-partum fully breastfeeding-

Exclusion Criteria:

* baby premature
* diabetes
* blood hypertension
* not breastfeeding or partial breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of infant weight, height and size of the tibial | women and children will be evaluated at time frame from day 42 through day 64 post-partum
  The study have the purpose to evaluate the infant weight, height and size of the tibial in infant who breastfeeding on demand exclusively and their mother were either users of a combined oral contraceptive, placebo, etonogestrel-releasing subdermal contraceptive implant or levonorgestrel-releasing intrauterine system. Additionally, pregnancy effectiveness and any adversse event will record in all groups of women.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Bahamondes, MD, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Bahamondes L, Bahamondes MV, Modesto W, Tilley IB, Magalhaes A, Pinto e Silva JL, Amaral E, Mishell DR Jr. Effect of hormonal contraceptives during breastfeeding on infant's milk ingestion and growth. Fertil Steril. 2013 Aug;100(2):445-50. doi: 10.1016/j.fertnstert.2013.03.039. Epub 2013 Apr 23. PMID 23623474